CLINICAL TRIAL: NCT05217511
Title: Effects of Neuromuscular Electrical Stimulation on Critically Ill Patients With Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, JinyanXing, Director, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DZH20220104
Record Dates: First submitted 2022-01-08; First posted 2022-02-01 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Respiratory Insufficiency Requiring Mechanical Ventilation
Keywords: Diaphragm ultrasound; Intercostal muscle ultrasound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMSE Group (Experimental): Neuromuscular Electrical Stimulation(NMES) group received consecutive daily sessions of electrical stimulation at specific points starting on the first day of randomization.The subjects also receive conventional physical therapy, which included gross motor therapy and respiratory therapy twice a day every day during their stay in the ICU.
  Interventions: Behavioral: Neuromuscular Electrical Stimulation
- CPT group (No Intervention): The subjects only receive conventional physical therapy, which included gross motor therapy and respiratory therapy twice a day every day during their stay in the ICU.

INTERVENTIONS:
Behavioral: Neuromuscular Electrical Stimulation — NMES was performed using a portable machine.The negative electrodes were placed in the motor points of the following muscles: chest muscles (pectoralis major muscle fibres) and rectus abdominis muscles bilaterally. A second (positive) electrode was positioned distally to the first, at a site close to the muscle that was being electrically stimulated, totalling 1 channel with 2 electrodes for each muscle . Each NMES session lasted 30 min. The following parameters were used: 50 Hz frequency, pulse duration 300 ms, rise time 1 s, stimulus time (ON) 3 s, decay time 1 s, and relaxation time (OFF) 10 s. Intensity was increased until muscle contraction was visible or could be identified through palpation. In conscious patients, intensity was adjusted according to their tolerance.
  Arms: NMSE Group

SUMMARY:
Up to 25% of patients who require mechanical ventilation (MV) more than seven days in the intensive care unit (ICU) develop muscle weakness, which comprises deep muscle weakness , including the respiratory muscles.Early active mobilization in ICU patients is a safe and viable strategy to prevent the physical problems caused by immobility. Neuromuscular electrical stimulation (NMES) is an alternative to mobilize and exercise because it does not require active patient participation and can be used on bedridden patients.No previous studies have shown whether training-specific respiratory muscles using an electrical stimulation can have overall benefits for ICU patients on MV.For this reason, the aim of this study was to evaluate, the effectiveness of the NMES therapy combined with early rehabilitation in the respiratory muscles of patients on MV.

ELIGIBILITY:
Inclusion Criteria:

* Prolonged MV(>72 h);
* Written informed consent was obtained from the patients or their relatives

Exclusion Criteria:

* Previous neuromuscular disease;
* Unrelieved pneumothorax, restricted diaphragmatic dyskinesia including abdominal high pressure, a large number of ascites
* Thoracic or diaphragmatic malformation;
* Local skin damage and infection;
* Indwelling a temporary or permanent pacemaker;
* Severe obesity(BMI>35 kg/m2)
* Various reasons (severe intestinal gas accumulation, structural abnormalities) lead to the failure of ultrasonic detection of diaphragm movement;
* Patients with an expected survival time of less than 7 days or with palliative care

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
diaphragmatic thickening fraction(DTF) | baseline,Day 3 of mechanical ventilation,Day 7 of mechanical ventilation,before extubation
  DTF shows varied thickness of the diaphragm at end-expiration and end-inspiration. Te maximum and minimum values of each breathing cycle were taken as the end-inspiratory diaphragm thickness (DTei) and the end-expiratory diaphragm thickness (DTee), respectively. DTF was calculated by DTF=(DTei DTee)/DTee 100%. Te values for 3 consecutive respiratory cycles were recorded and the average value was taken as the fnal value

SECONDARY OUTCOMES:
Parasternal Intercostal Muscle Ultrasound | baseline,Day 3 of mechanical ventilation,Day 7 of mechanical ventilation,before extubation
  A 10- to 15-MHz linear array transducer was positioned perpendicular to the anterior thorax surface in the longitudinal scan, at the level of the second right intercostal space, approximately 6 to 8 cm lateral to the sternal edge with a window visualizing the second and third ribs. . Using M-mode, the ultrasound beam was perpendicularly directed at the midsection of the muscle, where it is the thinnest at end-expiration. The thickness of the parasternal intercostal muscle was measured on frozen images at end expiration and at peak inspiration.

OTHER OUTCOMES:
ventilator-free days at 28 days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jinyan Xing, Dr., Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- Neuromuscular electrical stimulation, Qingdao, China